CLINICAL TRIAL: NCT03899376
Title: A Randomized Open-label Trial Comparing Acute Toxicity in Patients With Gynecological Cancer Treated With Adjuvant Conventional Versus VMAT Radiotherapy.
Brief Title: A Trial Comparing Acute Toxicity in Patients With Gynecological Cancer Treated With VMAT
Acronym: ATGCRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, David Cantu, Chief of clinical trial departament, National Institute of Cancerología
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 018/053/ICI CE/1309/18
Record Dates: First submitted 2019-03-01; First posted 2019-04-02 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Gynecologic Cancer
Keywords: Gynecological Cancer; Radiotherapy; VMAT; Toxicity
MeSH Terms: interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: a randomized open-label clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional radiotherapy (Active Comparator): patients with gynecological cancer treated with adjuvant conventional radiotherapy
  Interventions: Radiation: conventional radiotherapy
- Volumetric modulated arc therapy (Experimental): Patients with gynecological cancer treated with adjuvant VMAT radiotherapy
  Interventions: Radiation: Volumetric modulated arc therapy

INTERVENTIONS:
Radiation: Volumetric modulated arc therapy — VMAT therapy focuses on reducing the dose radiation in adjacent organs at risk
  Arms: Volumetric modulated arc therapy
Radiation: conventional radiotherapy — Radiotherapy focus on pelvis area
  Arms: Conventional radiotherapy

SUMMARY:
This is a randomized, controlled, open-label, prospective and longitudinal clinical trial. Rectal, intestinal and bladder EBRT-related toxicity will be assessed according to RTOG / EORTC scales at the first day of EBRT, during the 2nd, 3rd and 4th week of treatment, and 1, 3 and 6 months after the end of radiation treatment. The assessment of quality of life (QoL) will be measured by completing the questionnaire of the European Organization for Research and the Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-C30) version 3.0, in addition to specific QoL questionnaires for cervical and endometrial cancer respectively (EORTC QLQ-CX 24 and EORTC QLQ-EN24), previously validated in Mexican Spanish-speaking population, and which will be simultaneously applied with the RTOG / EORTC toxicity scales.

EXPECTED RESULTS AND PERSPECTIVES:

This trial aims to provide information about the feasibility of using a newer EBRT technique, as effective as conventional 3D-conformal radiation therapy (3D-CRT), but with less toxicity.

DETAILED DESCRIPTION:
BACKGROUND:

The standard of care in gynecological malignancies with high-risk features of recurrence following surgery is adjuvant external beam radiation therapy (EBRT) in the pelvic region, with or without concurrent chemotherapy (CT). This treatment modality offers higher local control and improves overall survival. EBRT has been associated with secondary effects due to toxicity such as cystitis, enteritis and proctitis which can compromise its effectiveness, patient´s quality of life and the interruption of the treatment. Newer EBRT techniques reduce the radiation dosis in normal tissues, with less toxicity. So far, there are no records of radiation-induced toxic effects in our population. The aim of this study is to evaluate the acute toxicity associated with pelvic postoperative EBRT using conventional or VMAT (RapidArc) technique in patients with gynecological cancer.

METHODOLOGY:

This is a randomized, controlled, open-label, prospective and longitudinal clinical trial. Rectal, intestinal and bladder EBRT-related toxicity will be assessed according to RTOG / EORTC scales at the first day of EBRT, during the 2nd, 3rd and 4th week of treatment, and 1, 3 and 6 months after the end of radiation treatment. The assessment of quality of life (QoL) will be measured by completing the questionnaire of the European Organization for Research and the Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-C30) version 3.0, in addition to specific QoL questionnaires for cervical and endometrial cancer respectively (EORTC QLQ-CX 24 and EORTC QLQ-EN24), previously validated in Mexican Spanish-speaking population, and which will be simultaneously applied with the RTOG / EORTC toxicity scales.

EXPECTED RESULTS AND PERSPECTIVES:

This trial aims to provide information about the feasibility of using a newer EBRT technique, as effective as conventional 3D-conformal radiation therapy (3D-CRT), but with less toxicity.

ELIGIBILITY:
Inclusion Criteria:

* patients with cervical or endometrial cancer with an indication of adjuvant radiotherapy after surgical treatment.

Exclusion Criteria:

* patients that reject to participate in the trial
* previous treatment with pelvic radiotherapy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patients with gynecological cancer with an indication of adjuvant radiotherapy after surgical treatment.
Enrollment: 80 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Acute Toxicity measured by toxicity scales | 1 year
  The acute toxicity will be measured, with RTOG acute radiation morbidity scoring criteria scale, this has four grades from 0 to 4, and higher values represent a worse outcome. The principal symptoms to evaluate are genitourinary and lower gastrointestinal.

SECONDARY OUTCOMES:
Quality of life measured by questionnaire | 1 year
  measured by completing the questionnaire of the European Organization for Research and the Treatment of Cancer Quality of Life Questionnaire C-30 (EORTC QLQ-C30) version 3.0, previously validated in Mexican Spanish-speaking population.
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items..
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

CONTACTS AND LOCATIONS:
Locations (1):
- David Cantu de Leon, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No